CLINICAL TRIAL: NCT03880006
Title: Leveraging Adaptive Implementation Strategies to Achieve Universal Coverage of Antiretroviral Treatment in Senegal
Brief Title: Universal Coverage of Antiretroviral Treatment in Senegal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); ENDA Sante, Senegal (Unknown); Ministry of Health, Senegal (Other Government); Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00007193
Record Dates: First submitted 2017-06-20; First posted 2019-03-19 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Case Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Participants assigned to the Senegalese standard of care treatment for people living with HIV.
- Case management (Experimental): Individuals in the intervention arm will receive Senegalese standard of care treatment for people living with HIV, and the case management intervention.
  Interventions: Behavioral: Case management

INTERVENTIONS:
Behavioral: Case management — Case management intervention is a multi-step process to coordinate care and provide a family-like support system for people living with HIV. Individuals are assigned to a specific case manager who will provide support throughout the study. The case management approach has five key components: 1) initial meeting between person living with HIV and case manager; 2) follow up meeting between case manager and participant; 3) biweekly automatic text messages sent to participant; 4) monthly phone calls from case manager; and 5) face-to-face meetings between case manager and participant every 6 months.
  Arms: Case management

SUMMARY:
Senegal plans a rapid scale up of HIV treatment for all people living with HIV, regardless of cluster of differentiation 4 (CD4) count or viral suppression. However, limited data exist on how to achieve sustained viral suppression outside of a controlled setting, and with significant barriers to effective antiretroviral therapy delivery, uptake, and adherence. The purpose of this study is to develop and assess the feasibility, fidelity, and cost-effectiveness of a universal coverage of Antiretroviral Treatment (ART) intervention among people living with HIV who are not virally suppressed in Dakar and Ziguinchor, Senegal.

DETAILED DESCRIPTION:
The overarching goal of this study is to assess the feasibility, fidelity, and cost-effectiveness of a universal coverage of Antiretroviral Treatment (ART) intervention among individuals living with HIV who are not virally suppressed in Dakar and Ziguinchor, Senegal. Specific aims and hypotheses are as follows:

Specific Aim 1: Compare the effectiveness and durability of (a) the existing Standard of Care (SOC) in Senegal versus (b) individual Case Management (CM) programs to achieve sustained viral suppression (SVS) among people living with HIV in Senegal.

Hypothesis 1: The null hypothesis is that standard of care and case management will be equally effective at achieving sustained viral suppression. The alternate hypothesis is that case management will be 30% more effective at sustained viral suppression at 12 months compared to standard of care.

Specific Aim 2: Determine the cost-effectiveness of the universal treatment approach using the CM intervention.

Hypothesis 1: A Case Management approach will be more cost-effective at achieving sustained viral suppression among people living with HIV (PLHIV) versus the existing standard of care in Senegal.

This study is a randomized controlled trial (RCT) that uses an effectiveness-implementation hybrid design to test the effectiveness and durability of CM interventions in achieving SVS among PLHIV who are not virally suppressed. CM vs. SOC approaches will be assessed using an individual-level RCT of case management to improve viral suppression of those living with HIV at 12 months compared to the Senegal SOC. While viral suppression will be a primary outcome of this intervention, significant attention will be given to the collection of service and implementation outcomes to assess both the SOC and CM.

Study sites will include two government HIV treatment facilities in Ziguinchor, and two in Dakar. Participant enrollment into the study will take place at the study sites, and study arms (SOC or CM) will be assigned through individual randomization at the clinic level. Notably, the HIV treatment facilities in this study are existing government facilities given the partnership between this study and the Ministry of Health (MOH) of Senegal.

Eligible participants recruited through the study site health facilities will go through the consent process in private rooms within the project office and complete a structured 1-hour interviewer-administered questionnaire, which will serve as the baseline assessment. Participants will be enrolled into the study, by trained study staff at a study site.

Baseline assessment of study participants will include a socio-behavioral questionnaire and biological testing. The baseline questionnaire will assess demographic characteristics, socioeconomic status, mobility and migration history, behavioral characteristics, health and HIV treatment history, and HIV acquisition risks.

Follow up will involve visits at 3, 6, 9, and 12 months after the first visit. Questionnaires will be administered at each visit. Questionnaires assessing behavioral characteristics, mental health, social support, and ART treatment adherence will be administered at 6 months, and 12 months.

Abbreviated questionnaires will be re-administered at 3 and 9 months though no biological assessments will be completed at these time points. The questionnaires leverage existing instruments that have detailed assessments engagement in ART services as well as enacted, perceived, and intersectional stigma. In addition, the investigators will use implementation indicators that explore measures of acceptability, fidelity, appropriateness, and routinization of the CM intervention.

Biological samples using either aliquots of serum or dried blood spots (DBS) will be taken at baseline, 6 months, and 12 months to support syphilis testing, HIV viral load, and other sexually transmitted infections (STIs). Biological testing taken at baseline and will include testing currently being implemented through the SOC, and testing conducted at the additional visits will be supported by the study. All participants will also have the opportunity to receive referrals for additional medical care as needed at the clinics in which the study sites are housed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Is mentally sound and capable of providing consent to participate
* Agrees to complete HIV and syphilis testing
* Speaks either French, Wolof or both
* Has provided informed consent to participate in the study
* Resident of Senegal for the past 3 months
* Intention to live in Dakar or Ziguinchor for the next 12 months
* Agrees to complete all required biological testing described in the consent form and receive results

Exclusion Criteria:

* Under 18 years of age
* Demonstrates mental incapacity, under the influence of substances, or any other illness preventing comprehension of the study procedures and informed consent
* Does not agree to complete all required biological testing described in the consent form or receive results
* Has not provided informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Viral suppression among study participants measured through biological samples using either aliquots of serum or dried blood spots (DBS). | Viral suppression at 12 months of follow up
  Biological samples using either aliquots of serum or dried blood spots will be taken at baseline, 6 months, and 12 months to support HIV viral load testing. Biological testing taken at baseline and will include testing currently being implemented through the SOC, and testing conducted at the additional visits will be supported by the study. All participants will also have the opportunity to receive referrals for additional medical care as needed at the clinics in which the study sites are housed.
  Sustained viral suppression is defines as quantitative viral load assessment with <1000 copies/ml at 12 months after initial randomization

SECONDARY OUTCOMES:
Loss-to-follow-up of study participation among study participants | Loss to follow up at 12 months
  Numbers and proportions of participants remaining engaged in the study will be measured through study visits every 3 months. Loss to follow up among participants in the existing Standard of Care study arm will be compared to the individual Case Management (CM) study arm to measure a difference in loss to follow up between the two study arms.
Acceptability of CM intervention among study participants through self-reported measure. | 12 months
  Acceptability of the CM intervention will be measured through self-reported measures collected through the social behavioral questionnaire. Acceptability measure is leveraged from the Society of Implementation Research Collaboration instrument review.
Cost-effectiveness of the universal treatment approach using the CM intervention | 12 months
  To determine the cost-effectiveness of the universal treatment approach using the CM intervention, we will perform a comprehensive costing of our study intervention, from the perspectives of both the healthcare system and the participants. Our costing methodology will follow World Health Organization (WHO) recommendations for cost-effectiveness analysis, with estimates of unit costs compared against WHO's CHOosing Interventions that are Cost-Effective (CHOICE) global estimates for countries in Senegal's region.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Baral, MD MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (4):
- Senegal (4):
  - Institut d'hygiene sociale / polyclinique, Dakar
  - Centre de sante Dominique, Pikine
  - Hopital regional de Ziguinchor, Ziguinchor
  - Hopital Silence de Ziguinchor, Ziguinchor

IPD SHARING:
Plan to Share IPD: No